CLINICAL TRIAL: NCT03285750
Title: Expression of GPR120 Receptor in Adipose Tissue of Type 2 Diabetic Subjects
Brief Title: Expression of G-protein Coupled Receptor 120 Receptor in Adipose Tissue of German Diabetes Center Cohort Subjects
Acronym: GPR120
Status: Completed | Type: Observational
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: GPR120 study
Record Dates: First submitted 2013-08-13; First posted 2017-09-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
Keywords: GPR120; Adipose tissue; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — SNP Genotyping of GPR120
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic group: Patients with recently diagnosed type 2 diabetes
- Controls: Age- and BMI-matched normoglycemic subjects

SUMMARY:
G-protein coupled receptor 120 (GPR120) is a G-protein-coupled receptor whose endogenous ligands have been identified as long-chain fatty acids. Recently, it has been shown that GPR120 expression in human adipose tissue is higher in obese than in lean individuals. Interestingly, a GPR120 deficient mouse model presents an unfavorable phenotype when fed a high-fat diet with obesity, glucose intolerance and fatty liver, characteristics also found in type 2 diabetes (T2D).

Moreover, in obese subjects, a single nucleotide polymorphism (R270H) has been identified that inhibits GPR120 signaling activity.

The investigators now want to investigate if GPR120 expression in adipose tissue may be altered in patients with T2D compared to non-diabetic subjects and might contribute to diabetes-associated metabolic changes. Additionally, the investigators want to assess the frequency of the R270H mutant in T2D.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus / normoglycemia
* BMI < 27,5 or > 30 kg/m2
* Age 20 - 69 years

Exclusion Criteria:

* severe chronic diseases
* anemia
* medication altering fatty acid metabolism

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with recently diagnosed type 2 diabetes (up to one year from diagnosis) and age- and weight-matched normoglycemic controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
GPR120 expression in adipose tissue | Expression measured at baseline (day 1)
  GPR expression is measured in adipose tissue of recently diagnosed type 2 diabetic patients and age- and BMI-matched normoglycemic controls

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany